CLINICAL TRIAL: NCT01452750
Title: A Phase 3, Multicenter, Randomized, Double-blind, AG-1749-controlled, Parallel-group, Comparison Study to Evaluate the Efficacy and Safety of TAK-438 (10 mg or 20 mg, Orally, Once Daily) for the Prevention of Recurrent Gastric or Duodenal Ulcers During Long-term Therapy of Non-steroidal Anti-inflammatory Drug (NSAID).
Brief Title: Efficacy and Safety of TAK-438 for the Prevention of Recurrent Gastric or Duodenal Ulcers During Therapy of Non-steroidal Anti-inflammatory Drug (NSAID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-438/CCT-301; U1111-1123-8722 (Registry Identifier: WHO); JapicCTI-111613 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-16; First posted 2011-10-17 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Gastric Ulcers; Duodenal Ulcers
Keywords: Drug Therapy
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-438 10 mg QD (Experimental)
  Interventions: Drug: TAK-438; Drug: Placebo
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438; Drug: Placebo
- Lansoprazole 15 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole; Drug: Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 10 mg tablets, orally, once daily for up to 24 weeks.
  Arms: TAK-438 10 mg QD
Drug: Placebo — Lansoprazole placebo-matching capsules, orally, once daily for up to 24 weeks.
  Arms: TAK-438 10 mg QD
Drug: TAK-438 — TAK-438 20 mg tablets, orally, once daily for up to 24 weeks.
  Arms: TAK-438 20 mg QD
Drug: Placebo — Lansoprazole placebo-matching capsules, orally, once daily for up to 24 weeks.
  Arms: TAK-438 20 mg QD
Drug: Lansoprazole — Lansoprazole 15 mg capsules, orally, once daily for up to 24 weeks.
  Other Names: AG-1749
  Arms: Lansoprazole 15 mg QD
Drug: Placebo — TAK-438 placebo-matching tablets, orally, once daily for up to 24 weeks.
  Arms: Lansoprazole 15 mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy of TAK-438, once daily (QD), compared to AG-1749 (Lansoprazole) in patients with a history of gastric or duodenal ulcer who require long-term therapy of non-steroidal anti-Inflammatory drug (NSAID).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who require continuous NSAID therapy during the treatment period with the study drug
2. Participants who have a history of ulcer in stomach or duodenum, endoscopically confirmed
3. Outpatient (including inpatient for examinations)

Exclusion Criteria:

1. Participants scheduled to change the type and dosage regimen of NSAID
2. Participants with ulcers or bleeding in stomach or duodenum, endoscopically confirmed
3. Participants with small intestine bleeding, large intestine bleeding, or gastrointestinal bleeding of unknown etiology
4. Participants who have a history of surgery which affects gastric acid secretion (e.g., resection of upper gastrointestinal tract, vagotomy) or who are scheduled to undergo such surgery
5. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders
6. Participants with a previous or current history of aspirin-induced asthma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of gastric or duodenal ulcer within 24 weeks | 24 weeks
  Mucosal defects with a white coating of 3 mm or larger will be determined as ulcers. Recurrence rate of gastric or duodenal ulcer within 24 weeks will be calculated for each treatment group.

SECONDARY OUTCOMES:
Recurrence rate of gastric or duodenal ulcer within 12 weeks | 12 weeks
Gastric mucosal injury | 24 Weeks
Duodenal mucosal injury | 24 weeks
Occurrence rate of hemorrhagic lesion in stomach or duodenum | 24 weeks
Time to recurrence of gastric or duodenal ulcer | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (102):
- Japan (102):
  - Kasugai-shi, Aichi-ken
  - Nagoya, Aichi-ken
  - Seto-shi, Aichi-ken
  - Akita, Akita
  - Funabashi-shi, Chiba
  - Ichihara-shi, Chiba
  - Nagareyama-shi, Chiba
  - Matsuyama, Ehime
  - Niihama-shi, Ehime
  - Saijo-shi, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Itoshima-shi, Fukuoka
  - Kitakyusyu-shi, Fukuoka
  - Munakata-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Tagawa-shi, Fukuoka
  - Yukuhashi-shi, Fukuoka
  - Fukushima, Fukushima
  - Koriyama-shi, Fukushima
  - Gifu, Gifu
  - Mebashi-shi, Gunma
  - Takasaki-shi, Gunma
  - Fukuyama-shi, Hiroshima
  - Hatsukaichi-shi, Hiroshima
  - Higashihirosima-shi, Hiroshima
  - Asahikawa-shi, Hokkaido
  - Hakodate-shi, Hokkaido
  - Obihiro-shi, Hokkaido
  - Sapporo, Hokkaido
  - Sunagawa-shi, Hokkaido
  - Tomakomai-shi, Hokkaido
  - Akashi-shi, Hyōgo
  - Himeji-shi, Hyōgo
  - Itami-shi, Hyōgo
  - Kako-gun, Hyōgo
  - Kato-shi, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Higashiibaragi-gun, Ibaragi
  - Koga-shi, Ibaragi
  - Mito, Ibaragi
  - Hitachi-shi, Ibaraki
  - Hakusan-shi, Ishikawa-ken
  - Komatsu-shi, Ishikawa-ken
  - Takamatsu, Kagawa-ken
  - Kamakura-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Uji-shi, Kyoto
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Matsumoto-shi, Nagano
  - Nagano, Nagano
  - Nagasaki, Nagasaki
  - Ikoma-shi, Nara
  - Nara, Nara
  - Nigata-shi, Niigata
  - Beppu-shi, Oita Prefecture
  - Ōita, Oita Prefecture
  - Yuhu-shi, Oita Prefecture
  - Kurashiki-shi, Okayama-ken
  - Higashiosaka-shi, Osaka
  - Moriguchi-shi, Osaka
  - Osaka, Osaka
  - Osakasayama-shi, Osaka
  - Tondabayashi-shi, Osaka
  - Ogi-shi, Saga-ken
  - Saga, Saga-ken
  - Ageo-shi, Saitama
  - Hiki-gun, Saitama
  - Kasukabe-shi, Saitama
  - Kumagaya-shi, Saitama
  - Saitama-shi, Saitama
  - Sayama-shi, Saitama
  - Toda-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Ōtsu, Shiga
  - Izumo-shi, Shimane
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Naruto-shi, Tokushima
  - Adachi-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Hachiouji-shi, Tokyo
  - Koto-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka-shi, Tokyo
  - Musashimurayama-shi, Tokyo
  - Nakano-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Sumida-ku, Tokyo
  - Yonago-shi, Tottori
  - Tonami-shi, Toyama
  - Toyama, Toyama
  - Shimonoseki-shi, Yamaguchi
  - Ube-shi, Yamaguchi

REFERENCES:
- [Derived] Mizokami Y, Oda K, Funao N, Nishimura A, Soen S, Kawai T, Ashida K, Sugano K. Vonoprazan prevents ulcer recurrence during long-term NSAID therapy: randomised, lansoprazole-controlled non-inferiority and single-blind extension study. Gut. 2018 Jun;67(6):1042-1051. doi: 10.1136/gutjnl-2017-314010. Epub 2017 Oct 7. PMID 28988197